CLINICAL TRIAL: NCT06787404
Title: Evaluation of Post-Induction Hypotension Treatment with PRAM Method Data in Gynecologic Oncology Cases
Brief Title: Evaluation of Post-Induction Hypotension Treatment with PRAM Method
Status: Active, not recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: E2-23-5996
Record Dates: First submitted 2024-12-09; First posted 2025-01-22 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Hypotension on Induction
Keywords: Post-induction Hypotension; PRAM; Ephedrine; Noradrenaline
MeSH Terms: interventions — Ephedrine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Ephedrine: When post-induction hypotension occurred patients were treated with 5 milligrams ephedrine in this group. If blood pressure does not reach desired levels, same dosage will be repeated 5 minutes later from administration. Maximum 3 doses will be applied and if hypotension ist persist the treatment will changed to rescue treatment.
  Interventions: Drug: Ephedrine
- Noradrenaline: When post-induction hypotension occurred patients were treated with 5 micrograms noradrenaline in this group. If blood pressure does not reach desired levels, same dosage will be repeated 5 minutes later from administration. Maximum 3 doses will be applied and if hypotension ist persist the treatment will changed to rescue treatment.
  Interventions: Drug: Noradrenalin

INTERVENTIONS:
Drug: Ephedrine — 5 milligrams of ephedrine will be applied when post-induction hypotension occured. After 3 doses, dose will be increased or changed to other treatment options.
  Other Names: Ephedrine Group
  Groups: Ephedrine
Drug: Noradrenalin — 5 micrograms of ephedrine will be applied when post-induction hypotension occured. After 3 doses, dose will be increased or changed to other treatment options.
  Other Names: Noradrenalin Group
  Groups: Noradrenaline

SUMMARY:
The goal of this observational study is to compare post-induction hypotension treatments with PRAM method in Gynecologic Oncological Cases. The goal of this observational study is to compare post-induction hypotension treatments with PRAM method in Gynecologic Oncological Cases.

DETAILED DESCRIPTION:
Post-induction hypotension is defined as hypotension that occurs within the first 20-30 minutes after general anesthesia induction or during the period between anesthesia induction and surgical incision. The global incidence rates are reported to be approximately 10.3%, with some studies indicating rates as high as 66.96%. Post-induction hypotension is associated with increased postoperative morbidity risks, such as acute kidney injury, transient tubular dysfunction, myocardial injury, and the need for postoperative intensive care. However, hypotension is a modifiable and preventable risk factor; its early detection and appropriate treatment can improve patient outcomes.

For this reason, investigators aimed to investigate the repeated dose requirements of alpha-adrenergic drugs, the recurrence of hypotension, and their effects on parameters observed via the MostCare monitor in patients undergoing major gynecologic oncologic surgeries during standard anesthesia induction and maintenance. This investigation focuses on patients experiencing a mean arterial pressure <65 mmHg or a >30% reduction in baseline systolic blood pressure within the first 30 minutes after induction or until surgical incision. Additionally, our secondary aim is to examine other parameters that may be associated with post-induction hypotension.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old
* Operated for Gynecologic Oncological reasons
* BMI<35

Exclusion Criteria:

* Refusal to participate in the study
* Additional spinal or epidural anesthesia
* Dementia patients from whom consent could not be obtained
* Atrial fibrillation with a rapid ventricular response
* Patients with difficult ventilation and/or difficult intubation
* Left ventricular ejection fraction (EF) below 30%
* Severe aortic valve stenosis
* Obesity (BMI >35)
* Chronic beta-blocker use

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Since our study is conducted on gynecologic oncology patients, all of our patients are women.
Study Population: The investigators choose Gynecological Oncology patients who will operated for gyno-oncological reasons
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
"Is there a difference in the need for repeated doses of treatments to reach the target blood pressure in patients who develop post-induction hypotension?" | First 30 minutes after anesthesia induction or time to skin incision
  When hypotension is occured, researchers applied two treatment (e.g. Ephedrine and Norepinephrine) and assessed how many hypotension episodes occured after treatment
"Is there a difference in the time to reach the target blood pressure after treatments in patients who develop post-induction hypotension?" | First 30 minutes after anesthesia induction or time to skin incision
  When hypotension is occured, researchers applied two treatment (e.g. Ephedrine and Norepinephrine) and assessed that is there a difference in the time to reach the target blood pressure after treatments

SECONDARY OUTCOMES:
Systemic vascular resistance (SVR) | First 30 minutes after anesthesia induction or time to skin incision
  To examine the effects of the applied treatments on the systemic vascular resistance from the PRAM method and compare them with each other.
Arterial Elastance (Ea) | First 30 minutes after anesthesia induction or time to skin incision
  To examine the effects of the applied treatments on the Ea from the PRAM method and compare them with each other.
Cardiac Output (CO) | First 30 minutes after anesthesia induction or time to skin incision
  To examine the effects of the applied treatments on the CO from the PRAM method and compare them with each other.
Stroke Volume (SV) | First 30 minutes after anesthesia induction or time to skin incision
  To examine the effects of the applied treatments on the SV from the PRAM method and compare them with each other.
Cardiac Cycle Efficiency (CCE) | First 30 minutes after anesthesia induction or time to skin incision
  To examine the effects of the applied treatments on the CCE from the PRAM method and compare them with each other.

CONTACTS AND LOCATIONS:
Overall Officials: Akgün E Şarer, Ass. Prof., Study Director — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent Şehir Hastanesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided